CLINICAL TRIAL: NCT02790138
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 4 Study to Evaluate the Efficacy and Safety of Entyvio (Vedolizumab IV) in the Treatment of Chronic Pouchitis (EARNEST)
Brief Title: A Study to Evaluate the Efficacy and Safety of Vedolizumab in the Treatment of Chronic Pouchitis
Acronym: EARNEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vedolizumab-4004; U1111-1171-0918 (Registry Identifier: WHO); 2015-003472-78 (EudraCT Number)
Record Dates: First submitted 2016-05-26; First posted 2016-06-03 (Estimated); Results first posted 2021-06-30 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Pouchitis
Keywords: Drug Therapy
MeSH Terms: conditions — Pouchitis | interventions — Ciprofloxacin; vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo IV (Placebo Comparator): Vedolizumab placebo-matching intravenous (IV) infusion, once at Day 1, Weeks 2, 6, 14, 22, and 30 along with ciprofloxacin 500 mg, tablet, orally twice daily up to Week 4.
  Interventions: Drug: Vedolizumab Placebo; Drug: Ciprofloxacin
- Vedolizumab IV 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, once at Day 1, Weeks 2, 6, 14, 22, and 30 along with ciprofloxacin 500 mg, tablet, orally twice daily up to Week 4.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab Placebo — Vedolizumab placebo-matching IV infusion
  Arms: Placebo IV
Drug: Ciprofloxacin — Ciprofloxacin tablets
  Arms: Placebo IV
Drug: Vedolizumab — Vedolizumab IV infusion
  Other Names: Entyvio; MLN0002 IV; Kynteles
  Arms: Vedolizumab IV 300 mg

SUMMARY:
The purpose of this study is to compare the efficacy of vedolizumab intravenous (IV) and placebo in terms of the percentage of participants with chronic or recurrent pouchitis achieving clinically relevant remission.

DETAILED DESCRIPTION:
Vedolizumab is being tested to treat people who have chronic pouchitis. This study will look at the healing of inflammation of ileal pouch in people who take vedolizumab as compared to those receiving a matching placebo. The study will enroll approximately 110 patients. Participants will be randomly assigned to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Vedolizumab 300 mg IV
* Placebo IV

All participants will receive an intravenous infusion at Day 1, Weeks 2, 6, 14, 22, and 30 along with concomitant antibiotic treatment with ciprofloxacin 500 mg twice daily through Week 4.

This multicenter trial will be conducted in North America and Europe. The overall time to participate in treatment and efficacy assessment of this study is 34 weeks. Participants will make multiple visits to the clinic, plus a final visit 18 weeks after the last dose of study drug for a safety follow-up assessment (up to Week 48). Participants will also participate in a long-term follow-up, by phone after the last dose of study drug up to Week 56.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a history of ileal pouch anal anastomosis (IPAA) for ulcerative colitis (UC) completed at least 1 year prior to the Day 1 (Randomization) Visit.
4. Has pouchitis that is chronic or recurrent, defined by an modified pouchitis disease activity index (mPDAI) score ≥5 assessed as average from 3 days immediately prior to the Baseline endoscopy and a minimum endoscopic subscore of 2 (outside the staple or suture line) with either (a) ≥3 recurrent episodes within 1 year prior to the Screening Period treated with ≥2 weeks of antibiotic or other prescription therapy, or (b) requiring maintenance antibiotic therapy taken continuously for ≥4 weeks immediately prior to the Baseline Endoscopy Visit.
5. Agrees to take ciprofloxacin (500 mg twice daily) on Day 1 and through Week 4, regardless of the previous treatment and to stop any previous antibiotic therapy on Day 1 of the study (additional courses of antibiotics will be allowed, as needed, for flares after Week 14).
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use a barrier method of contraception (e.g., condom with spermicide) from signing of informed consent throughout the duration of the study and for 18 weeks after last dose. The female partner of a male participant should also be advised to use a highly effective method of contraception.
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use a highly effective method of contraception from signing of informed consent throughout the duration of the study and for 18 weeks after last dose.

Exclusion Criteria:

Gastrointestinal Exclusion Criteria

1. Has Crohn's disease (CD), or CD of the pouch.
2. Has irritable pouch syndrome (IPS).
3. Has isolated or predominant cuffitis.
4. Has mechanical complications of the pouch (e.g., pouch stricture or pouch fistula).
5. Currently requires or has a planned surgical intervention for UC during the study.
6. Has diverting stoma.

Infectious Disease Exclusion Criteria 1. Has evidence of an active infection (e.g., sepsis, cytomegalovirus, or listeriosis) during Screening.

2. Has active or latent tuberculosis (TB), regardless of treatment history, as evidenced by any of the following:

1. A diagnostic TB test performed within 30 days of Screening or during the Screening Period that is positive, as defined by:

   1. A positive QuantiFERON test or 2 successive indeterminate QuantiFERON tests. OR
   2. A tuberculin skin test reaction ≥10 mm (≥5 mm in participants receiving the equivalent of >15 mg/day prednisone).

      OR
2. Chest X-ray within 3 months prior to Day 1 that is suspicious for pulmonary TB, and a positive or 2 successive indeterminate QuantiFERON test within 30 days prior to Screening or during the Screening Period.

   3. Has chronic hepatitis B virus (HBV) infection* or chronic hepatitis C virus (HCV) infection** or a known history of human immunodeficiency virus (HIV) infection (or is found to be seropositive at Screening) or participant is immunodeficient (e.g., due to organ transplantation, history of common variable immunodeficiency, etc).

   * Participants who are positive for hepatitis B virus surface antigen (HBsAg) will be excluded. For participants who are negative for HBsAg but are positive for either surface antibodies and/or core antibodies, HBV Deoxyribonucleic acid (DNA) polymerase chain reaction will be performed and if any test result meets or exceeds detection sensitivity, the participant will be excluded.
   * If participant is HCV antibody positive, then a viral load test will be performed. If the viral load test is positive then the participant will be excluded.

     4. Has evidence of active infection with Clostridium (C) difficile during Screening (to be confirmed by laboratory test)

   General Exclusion Criteria
   1. Has any prior exposure to vedolizumab, natalizumab, efalizumab, rituximab, etrolizumab, or anti-mucosal addressin cell adhesion molecule-1 (MAdCAM-1) therapy.
   2. Has a history of hypersensitivity or allergies to vedolizumab or its components.
   3. Has allergies to and/or contraindications for ciprofloxacin, a history of tendon disorders related to quinolone administration and/or glucose-6-phosphate dehydrogenase (G6PD) deficiency. Further conditions requiring precautions for use of ciprofloxacin have to be considered based on local prescribing information.
   4. Is taking, has taken, or is required to take any excluded medications.
   5. Has received any investigational or approved biologic or biosimilar agent within 60 days prior to Randomization.
   6. Has received an investigational nonbiologic therapy within 30 days prior to Randomization.
   7. Has received an approved nonbiologic therapy (including 5-aminosalicylate [5-ASA], corticosteroid, azathioprine, 6-mercaptopurine [6-MP], etc.) in an investigational protocol within 30 days prior to Randomization.
   8. Has received any live vaccinations within 30 days prior to randomization.
   9. Has a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist at Screening.
   10. Has had a kidney, heart, or lung transplant.
   11. Has a history of malignancy, except for the following: adequately-treated non-metastatic basal cell skin cancer; squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to the Screening visit; and history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to Screening. Participants with a remote history of malignancy (e.g., >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with the sponsor on a case-by-case basis prior to enrollment.
   12. Has a history of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, demyelinating, or neurodegenerative disease.
   13. Has conditions, which in the opinion of the investigator, may interfere with the participant's ability to comply with the study procedures.
   14. Has any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal (GI), genitourinary, hematological, coagulation, immunological, endocrine/metabolic, neurologic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise participant safety.
   15. Has any of the following laboratory abnormalities during the Screening Period:

   <!-- -->

   1. Hemoglobin level <8 g/dL.
   2. White blood cell (WBC) count <3 × 10^9/L.
   3. Lymphocyte count <0.5 × 10^9/L.
   4. Platelet count <100 × 10^9/L or >1200 × 10^9/L.
   5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × the upper limit of normal (ULN).
   6. Alkaline phosphatase >3 × ULN.
   7. Serum creatinine >2 × ULN.

   16. If female, the participant is pregnant or lactating or intending to become pregnant or nurse before, during, or within 18 weeks after the last dose of study medication; or intending to donate ova during such time period.

   17. If male, the participant intends to donate sperm or father a child during the course of this study or for 18 weeks after the last dose of study medication.

   18. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.

   19. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (34):
- United States (10):
  - University of Chicago Medical Center, Chicago, Illinois
  - Northshore University HealthSystem, Evanston, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina GI, Chapel Hill, North Carolina
  - Carolinas HealthCare System Digestive Health, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Digestive Disease Consultants, Southlake, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
- UZ Leuven - University Hospital Gasthuisberg, Leuven, Belgium
- Canada (3):
  - GIRI (GI Research Institute), Vancouver, British Columbia
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
- France (4):
  - CHU de Rennes - Hopital de Pontchaillou, Rennes
  - CHU Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - CHU de Toulouse - Hopital Rangueil, Toulouse
  - CHRU Nancy Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Charite Universitatsmedizin Berlin -Campus Virchow Klinikum, Berlin
  - Asklepios Hospital Hamburg - West, Hamburg
  - Praxis fuer Gastroenterologie, Drs. Ehehalt/ Helmstaedter, Heidelberg
  - Universitatsklinikum Jena, Jena
  - Klinikum Mannheim GmbH Universitaetsklinikum, Mannheim
- Italy (4):
  - Azienda Ospedaliera S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera di Padova, Padua
  - Policlinico Gemelli, Rome
  - Istituto Clinico Humanitas IRCCS, Rozzano
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Maastricht University Medical Center, Maastricht
- Spain (2):
  - Hospital Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario y Politecnico La Fe, Valencia
- United Kingdom (3):
  - St. Mark's Hospital, Harrow
  - Royal London Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Jairath V, Feagan BG, Silverberg MS, Danese S, Gionchetti P, Lowenberg M, Bressler B, Ferrante M, Hart A, Lindner D, Escher A, Jones S, Shen B, Travis S. Mucosal Healing With Vedolizumab in Patients With Chronic Pouchitis: EARNEST, a Randomized, Double-Blind, Placebo-Controlled Trial. Clin Gastroenterol Hepatol. 2025 Feb;23(2):321-330.e3. doi: 10.1016/j.cgh.2024.06.037. Epub 2024 Jul 16. PMID 39025255
- [Derived] Travis S, Silverberg MS, Danese S, Gionchetti P, Lowenberg M, Jairath V, Feagan BG, Bressler B, Ferrante M, Hart A, Lindner D, Escher A, Jones S, Shen B; EARNEST Study Group. Vedolizumab for the Treatment of Chronic Pouchitis. N Engl J Med. 2023 Mar 30;388(13):1191-1200. doi: 10.1056/NEJMoa2208450. PMID 36988594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 31 investigative sites in Canada, United States, Belgium, France, Germany, Italy, Netherlands, Spain, and United Kingdom from 12 October 2016 to 2 February 2021.
Pre-assignment Details: Participants with a diagnosis of chronic or recurrent pouchitis were enrolled in a 1:1 ratio to receive placebo IV or vedolizumab IV 300 mg.
Groups:
- Placebo IV: Vedolizumab placebo-matching IV infusion, once at Day 1, Weeks 2, 6, 14, 22, and 30 along with ciprofloxacin 500 mg, tablet, orally twice daily up to Week 4.
Period: Overall Study
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Started | 51 | 51
Completed | 30 | 32
Not Completed | 21 | 19
Not completed — Adverse Event | 5 | 2
Not completed — Significant Protocol Deviation | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Voluntary Withdrawal | 8 | 9
Not completed — Lack of Efficacy | 6 | 7
Not completed — Reason not Specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study medication, as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo IV | Vedolizumab IV 300 mg | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (13.48) | 40.8 (11.32) | 41.9 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 38 | 32 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 40 | 39 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 42 | 44 | 86
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 7 | 9 | 16
  United States | 11 | 12 | 23
  Belgium | 6 | 1 | 7
  France | 2 | 5 | 7
  Germany | 1 | 2 | 3
  Italy | 10 | 10 | 20
  Netherlands | 6 | 4 | 10
  Spain | 1 | 0 | 1
  United Kingdom | 7 | 8 | 15
Height [Mean (Standard Deviation); unit: cm] | 175.3 (9.10) | 172.4 (10.79) | 173.8 (10.04)
Weight [Mean (Standard Deviation); unit: kg] | 79.60 (19.115) | 72.13 (17.588) | 75.87 (18.658)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = weight (kg)/[height (m)^2
  kg/m^2 | 25.74 (5.125) | 24.13 (4.891) | 24.93 (5.049)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Chronic or Recurrent Pouchitis Achieving Clinically Relevant Remission at Week 14
Description: Clinically relevant remission is defined as modified Pouchitis Disease Activity Index (mPDAI) score <5 and a reduction of mPDAI score by ≥2 points from Baseline. The 12-point mPDAI score is calculated as a sum of from two 6-point subscales, where 0 = best and 12 = worst.: 1) Clinical Symptoms: Stool Frequency (0=usual to postoperative stool frequency to 2=three or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever [temperature >37.8 degrees C] (0=Absent and 1=Present) for a clinical symptoms subscore of 0 (best) to 6 (worse); 2) Endoscopic Inflammation Findings: Edema, Granularity, Friability, Loss of vascular pattern, Mucous exudates and Ulcerations. Each item is scored on a scale of 0=not present to 1=present summed up to an endoscopic subscore ranging from 0 (best) to 6 (worst) where higher scores indicate more severe disease.
Time Frame: Week 14
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study medication, as randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Number analyzed (Participants) | 51 | 51
percentage of participants | 9.8 [3.3 to 21.4] | 31.4 [19.1 to 45.9]
Statistical Analysis 1: Comparison: Placebo IV vs Vedolizumab IV 300 mg; The Placebo IV and Vedolizumab IV 300 mg groups were analyzed using Fisher's Exact Test at Week 14; Test type: Superiority; p = 0.013, Fisher's Exact Test — The significance level was 0.05; Percentage Difference = 21.6, 95% CI 2-sided [4.9 to 37.5]

2. Secondary Outcome: Percentage of Participants With Chronic or Recurrent Pouchitis Achieving Clinically Relevant Remission at Week 34
Description: Clinically relevant remission is defined as mPDAI score <5 and a reduction of mPDAI score by ≥2 points from Baseline. The 12-point mPDAI score is calculated as a sum of from two 6-point subscales, where 0 = best and 12 = worst.: 1) Clinical Symptoms: Stool Frequency (0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever [temperature >37.8 degrees C] (0=Absent and 1=Present) for a clinical symptoms subscore of 0 (best) to 6 (worse); 2) Endoscopic Inflammation Findings: Edema, Granularity, Friability, Loss of vascular pattern, Mucous exudates and Ulcerations. Each item is scored on a scale of 0=not present to 1=present summed up to an endoscopic subscore ranging from 0 (best) to 6 (worst) where higher scores indicate more severe disease.
Time Frame: Week 34
Population: FAS included all randomized participants who received at least 1 dose of study medication, as randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Number analyzed (Participants) | 51 | 51
percentage of participants | 17.6 [8.4 to 30.9] | 35.3 [22.4 to 49.9]
Statistical Analysis 1: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Test type: Superiority; p = 0.043, Chi-squared Test — No multiplicity adjustment for inferential testing for secondary endpoints was preplanned, p-values from these tests are presented as nominal p-values. The significance level was 0.05; Percentage Difference = 17.6, 95% CI 2-sided [0.3 to 35.1]

3. Secondary Outcome: Percentage of Participants Achieving Pouchitis Disease Activity Index (PDAI) Remission at Weeks 14 and 34
Description: PDAI remission is PDAI score <7 and a reduction of PDAI score by ≥3 points from Baseline. The 18-point PDAI score is calculated as a sum of three 6-point scales with total possible subscore of 0 (best) to 6 (worse) and possible total score of 0 (best) to 18 (worse):1)Clinical Symptoms:Stool Frequency(0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual);Rectal bleeding(0=None or rare,1=Present daily);Fecal urgency/abdominal cramps(0=None to 2=Usual),Fever[temperature>37.8 degrees C](0=Absent,1=Present);2)Endoscopic Inflammation:Edema,Granularity,Friability,Loss of vascular pattern,Mucous exudates,Ulcerations. Each item is scored on scale of 0=not present to 1=present summed up to an endoscopic subscore ranging from 0(best) to 6(worst);3) Acute Histologic Inflammation:Polymorphic nuclear leukocyte infiltration(0=None to 3=Severe plus crypt abscess),Ulceration per low power field[mean](0=0% to 3=>50%) where higher scores indicate more severe disease.
Time Frame: Weeks 14 and 34
Population: FAS included all randomized participants who received at least 1 dose of study medication, as randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Number analyzed (Participants) | 51 | 51
percentage of participants
  Week 14 | 9.8 [3.3 to 21.4] | 35.3 [22.4 to 49.9]
  Week 34 | 17.6 [8.4 to 30.9] | 37.3 [24.1 to 51.9]
Statistical Analysis 1: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Week 14; Test type: Superiority; p = 0.004, Fisher's Exact Test — [p-value comment as in outcome 2, analysis 1]; Percentage Difference = 25.5, 95% CI 2-sided [8.0 to 41.4]
Statistical Analysis 2: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Week 34; Test type: Superiority; p = 0.027, Chi-squared Test — [p-value comment as in outcome 2, analysis 1]; Percentage Difference = 19.6, 95% CI 2-sided [1.9 to 37.0]

4. Secondary Outcome: Time to PDAI Remission
Description: Time to remission-time in days from start of treatment to PDAI Remission(PDAI score <7 and decrease in PDAI score ≥3 points from Baseline).18-point PDAI score-calculated as sum of 3, 6-point scales with total possible subscore of 0(best) to 6(worse) and possible total score of 0(best)to18(worse):1)Clinical Symptoms:Stool Frequency(0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual);Rectal bleeding(0=None or rare,1=Present daily);Fecal urgency/abdominal cramps(0=None to 2=Usual),Fever[temperature>37.8 degrees C](0=Absent,1=Present);2)Endoscopic Inflammation:Edema,Granularity,Friability,Loss of vascular pattern,Mucous exudates,Ulcerations.Each item is scored on scale of 0=not present to 1=present summed up to an endoscopic subscore=0(best) to 6(worst);3)Acute Histologic Inflammation:Polymorphic nuclear leukocyte infiltration(0=None to 3=Severe plus crypt abscess),Ulceration per low power field[mean](0=0% to 3=>50%),higher scores=more severe disease.
Time Frame: Baseline up to Week 34
Population: FAS included all randomized participants who received at least 1 dose of study medication, as randomized.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Number analyzed (Participants) | 51 | 50
days | NA [NA to NA] — Median and 95% Confidence Interval (CI) was not estimated due to the low number of participants with events. | 239.0 [101.0 to NA] — Upper limit of 95% CI was not estimated due do the low number of participants with events.
Statistical Analysis 1: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Test type: Superiority; Hazard Ratio (HR) = 3.95, 95% CI 2-sided [1.7 to 9.4] — Hazard ratio for achieving PDAI remission

5. Secondary Outcome: Percentage of Participants Achieving a Partial mPDAI Response at Weeks 14 and 34
Description: Partial mPDAI response is defined as a reduction in mPDAI score by ≥2 points from Baseline. The 12-point mPDAI score is calculated as a sum of from two 6-point subscales, where 0 = best and 12 = worst:1) Clinical Symptoms: Stool Frequency (0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever [temperature >37.8 degrees C] (0=Absent and 1=Present) for a clinical symptoms subscore of 0 (best) to 6 (worse); 2) Endoscopic Inflammation Findings: Edema, Granularity, Friability, Loss of vascular pattern, Mucous exudates and Ulcerations. Each item is scored on a scale of 0=not present to 1=present summed up to an endoscopic subscore ranging from 0 (best) to 6 (worst) where higher scores indicate more severe disease. Last observation carried forward (LOCF) method was used for analyses.
Time Frame: Weeks 14 and 34
Population: FAS included all randomized participants who received at least 1 dose of study medication, as randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Number analyzed (Participants) | 51 | 51
percentage of participants
  Week 14 | 33.3 [20.8 to 47.9] | 62.7 [48.1 to 75.9]
  Week 34 | 29.4 [17.5 to 43.8] | 51.0 [36.6 to 65.2]
Statistical Analysis 1: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Week 14; Test type: Superiority; p = 0.003, Chi-squared Test — [p-value comment as in outcome 2, analysis 1]; Percentage Difference = 29.4, 95% CI 2-sided [8.0 to 47.6]
Statistical Analysis 2: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Week 34; Test type: Superiority; p = 0.026, Chi-squared Test — [p-value comment as in outcome 2, analysis 1]; Percentage Difference = 21.6, 95% CI 2-sided [1.9 to 39.8]

6. Secondary Outcome: Change From Baseline in PDAI Endoscopic Inflammation Subscore at Weeks 14 and 34
Description: The PDAI Endoscopic Inflammation subscore is a sum of scores from findings for Edema, Granularity, Friability, Loss of vascular pattern, Mucous exudates, and Ulcerations, each scored on 0=not present to 1=present scale summed up to a subscore ranging from 0 (best) to 6 (worse) where higher scores = more severe disease. A negative change from Baseline indicates improvement. LOCF method was used for analyses.
Time Frame: Baseline up to Weeks 14 and 34
Population: FAS included all randomized participants who received at least 1 dose of study medication, as randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Number analyzed (Participants) | 51 | 51
score on a scale
  Baseline | 4.5 (1.36) | 4.6 (1.15)
  Change from Baseline at Week 14 | -0.2 (1.36) | -1.1 (1.59)
  Change from Baseline at Week 34 | -0.6 (1.86) | -1.2 (1.87)
Statistical Analysis 1: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 14; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; P-value is from Wilcoxon Rank-sum Test comparing change from Baseline to relevant visits.Wilcoxon-Mann-Whitney odds estimator,95% CI are presented; Odds Estimator = 2.02, 95% CI 2-sided [1.11 to 2.93]
Statistical Analysis 2: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 34; Test type: Superiority; p = 0.020, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.71, 95% CI 2-sided [0.92 to 2.49]

7. Secondary Outcome: Change From Baseline in PDAI Acute Histologic Inflammation Subscore at Weeks 14 and 34
Description: The PDAI Acute Histologic Inflammation subscore is a sum score from findings for Polymorphic nuclear leukocyte infiltration (0=None to 3=Severe plus crypt abscess), and Ulceration per low power field [mean] (0=0% to 3= >50%) summed up to a subscore ranging from 0 (best) to 6 (worse) where higher scores = more severe disease. A negative change from Baseline indicates improvement. LOCF method was used for analyses.
Time Frame: Baseline up to Weeks 14 and 34
Population: FAS included all randomized participants who received at least 1 dose of study medication, as randomized. Overall number analyzed are the number of participants with data evaluable for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Number analyzed (Participants) | 51 | 50
score on a scale
  Baseline | 2.6 (1.39) | 2.5 (1.42)
  Change from Baseline at Week 14 | -0.1 (1.33) | -0.4 (1.98)
  Change from Baseline at Week 34 | -0.2 (1.52) | -0.2 (2.03)
Statistical Analysis 1: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 14; Test type: Superiority; p = 0.191, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.34, 95% CI 2-sided [0.74 to 1.94]
Statistical Analysis 2: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 34; Test type: Superiority; p = 0.766, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.07, 95% CI 2-sided [0.60 to 1.54]

8. Secondary Outcome: Change From Baseline in Total PDAI Score at Weeks 14 and 34
Description: The 18-point PDAI score is calculated as a sum of three 6-point scales with total possible subscore of 0 (best) to 6 (worse) and possible total score of 0 (best) to 18 (worse):1)Clinical Symptoms:Stool Frequency(0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual);Rectal bleeding(0=None or rare,1=Present daily);Fecal urgency/abdominal cramps(0=None to 2=Usual),Fever[temperature>37.8 degrees C](0=Absent,1=Present);2)Endoscopic Inflammation:Edema,Granularity,Friability,Loss of vascular pattern,Mucous exudates,Ulcerations. Each item is scored on scale of 0=not present to 1=present summed up to an endoscopic subscore ranging from 0(best) to 6(worst);3)Acute Histologic Inflammation:Polymorphic nuclear leukocyte infiltration(0=None to 3=Severe plus crypt abscess),Ulceration per low power field[mean](0=0% to 3=>50%) where higher scores=more severe disease. A negative change from Baseline indicates improvement. LOCF method was used for analyses.
Time Frame: Baseline up to Weeks 14 and 34
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Number analyzed (Participants) | 51 | 50
score on a scale
  Baseline | 10.5 (2.48) | 10.5 (2.20)
  Change from Baseline at Week 14 | -1.3 (2.68) | -2.7 (3.86)
  Change from Baseline at Week 34 | -1.6 (3.41) | -2.9 (3.93)
Statistical Analysis 1: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 14; Test type: Superiority; p = 0.055, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.57, 95% CI 2-sided [0.83 to 2.31]
Statistical Analysis 2: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 34; Test type: Superiority; p = 0.095, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.48, 95% CI 2-sided [0.79 to 2.16]

9. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Weeks 14, 22, and 34
Description: The IBDQ is an instrument used to assess quality of life in adult participants with inflammatory bowel disease (IBD). It includes 32 questions on 4 domains of Health-Related Quality-of-Life (HRQOL): Bowel Systems (10 items), Emotional Function (12 items), Social Function (5 items), and Systemic Function (5 items). Participants are asked to recall symptoms and quality of life from the last 2 weeks and rate each item on a 7-point Likert scale (1=worst to 7=best). A total IBDQ score is calculated by summing the scores from each domain; the total IBDQ score ranges from 32 to 224, with lower scores reflecting worse HRQOL. A negative change from Baseline indicates worsening. LOCF method was used for analyses.
Time Frame: Baseline up to Weeks 14, 22, and 34
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Number analyzed (Participants) | 50 | 51
score on a scale
  Baseline | 131.5 (30.78) | 137.9 (33.53)
  Change from Baseline at Week 14 | 14.6 (26.67) | 18.3 (29.20)
  Change from Baseline at Week 22 | 16.0 (29.12) | 21.3 (31.28)
  Change from Baseline at Week 34 | 10.4 (25.98) | 24.4 (34.21)
Statistical Analysis 1: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 14; Test type: Superiority; p = 0.575, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.14, 95% CI 2-sided [0.61 to 1.67]
Statistical Analysis 2: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 22; Test type: Superiority; p = 0.403, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.21, 95% CI 2-sided [0.65 to 1.78]
Statistical Analysis 3: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 34; Test type: Superiority; p = 0.047, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.60, 95% CI 2-sided [0.85 to 2.34]

10. Secondary Outcome: Change From Baseline in Cleveland Global Quality of Life (CGQL) at Weeks 14, 22, and 34
Description: The CGQL (Fazio score) is a quality-of-life indicator specifically for participants with ileal pouch-anal anastomosis. Participants rate 3 items (current quality of life, current quality of health, and current energy level), each on a scale of 0 to 10 (0=worst; 10=best). The scores are added, and the final CGQL utility score is obtained by dividing this result by 30. The total score ranges from 0 (worst) to 1 (best) where lower scores indicate less quality of life. A negative change from Baseline indicates worsening. LOCF method was used for analyses.
Time Frame: Baseline up to Weeks 14, 22, and 34
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
Number analyzed (Participants) | 49 | 50
score on a scale
  Baseline | 0.522 (0.1953) | 0.556 (0.1626)
  Change from Baseline at Week 14 | 0.051 (0.1518) | 0.088 (0.1715)
  Change from Baseline at Week 22 | 0.073 (0.1491) | 0.093 (0.1648)
  Change from Baseline at Week 34 | 0.056 (0.1544) | 0.083 (0.1831)
Statistical Analysis 1: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 14; Test type: Superiority; p = 0.119, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.44, 95% CI 2-sided [0.77 to 2.12]
Statistical Analysis 2: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 22; Test type: Superiority; p = 0.542, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.15, 95% CI 2-sided [0.62 to 1.69]
Statistical Analysis 3: Comparison: Placebo IV vs Vedolizumab IV 300 mg; Change from Baseline at Week 34; Test type: Superiority; p = 0.404, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 6, analysis 1]; Odds Estimator = 1.22, 95% CI 2-sided [0.65 to 1.78]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 18 weeks after last dose (Up to 50 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo IV | Vedolizumab IV 300 mg
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 4/51 | 3/51
Other Adverse Events (participants affected / at risk) | 35/51 | 42/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo IV (N=51) | Vedolizumab IV 300 mg (N=51)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Pouchitis (Gastrointestinal disorders) | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo IV (N=51) | Vedolizumab IV 300 mg (N=51)
Pouchitis (Gastrointestinal disorders) | 20 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 7
Headache (Nervous system disorders) | 3 | 10
Nasopharyngitis (Infections and infestations) | 6 | 6
Nausea (Gastrointestinal disorders) | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Frequent bowel movements (Gastrointestinal disorders) | 2 | 4
Influenza (Infections and infestations) | 1 | 4
Gastroenteritis (Infections and infestations) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT02790138/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT02790138/SAP_001.pdf